CLINICAL TRIAL: NCT01432132
Title: Mirror Grant - Toward an Understanding of Body Image Adaptation Following Surgical Treatment for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-0558
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Body Image Adaptation; Post surgical body image; Audio-recorded interview; Questionnaire; Survey
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Head & Neck Patients: Patients undergoing surgical treatment for head and neck cancer.
  Interventions: Behavioral: Interview; Behavioral: Questionnaire
- Clinicians: Clinical staff who care for head and neck surgical participants during active treatment.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Face-to-face audio recorded interview. It should take about 1 hour to complete.
Behavioral: Questionnaire — Questionnaire about demographic information such as age and ethnicity.
  Other Names: Survey
  Groups: Head & Neck Patients

SUMMARY:
The goal of this research study is to understand how patients adjust to appearance and body image changes after surgery for head and neck cancer.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will take part in a face-to-face interview with the study staff. It should take about 1 hour to complete. You will also be asked to complete a questionnaire about your demographic information such as age and ethnicity. The interview will be done in a private research area and will be audio-recorded.

The researchers are interested in learning more about your experience of adjusting to the changes in your appearance after your surgery for head and neck cancer. You may be asked to look in a mirror and describe what you see.

If you ask for another interview, or if the interviewer would like your information made more clear, you will be scheduled for a second interview. You will be provided with an early summary of your interview, and you will be able to provide feedback over the phone or in writing on the accuracy of the information and the conclusions.

Identifying information will be removed from all data collected using participant numbers kept separately from consent forms and shared only among approved research staff. Names and other identifying information will be deleted from transcripts (write-ups of the interviews) after the first review for accuracy. Interview transcripts will be kept in locked file cabinets at MD Anderson for 3 years and can be looked at only by the study chair and staff. Recorded interviews will be destroyed 3 years after the study results are published.

This is an investigational study.

Up to 20 patients and 15 healthcare providers will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. English speaking
3. For patients: Within 6 weeks of undergoing surgical resection for a tumor in the head and neck region, or within 1-3 years from such surgery.
4. For providers: Inpatient clinical staff (i.e. surgeons, nurses, nursing assistants, physical therapists) who care for surgically treated head and neck cancer patients during acute postoperative recovery, and/or outpatient clinical staff (i.e. nurses, physician assistants) who care for these patients throughout active treatment and into the period of survivorship.
5. For providers: Having worked with surgically treated head and neck cancer patients for at least one year.

Exclusion Criteria:

1) For patients: cognitive impairment documented in their medical record (e.g. delirium, dementia) impeding the ability to offer a narrative of his/her experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from the Head and Neck Center at MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Patients' Body Image Adaptation (Interviews) | Study period 2 years to complete face-to-face interviews
  Patients' experiences of viewing themselves in the mirror immediately after surgical treatment for head and neck cancer. Descriptive information derived from 1 hour face-to-face interviews with qualitative methodology using Grounded Theory design and methods with use of constant comparative technique and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C. Fingeret, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org